CLINICAL TRIAL: NCT00394758
Title: Comparison of Surgical Procedures in Vulvar and Vaginal Dysplasias
Brief Title: A Randomized Trial of Surgical Treatments for Vulvar and Vaginal Dysplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE 4804
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Vulvar Dysplasia; Vaginal Dysplasia
Keywords: ultrasonic surgical aspiration; CO2 laser surgery; vulvar dysplasia; vaginal dysplasia; recurrence
MeSH Terms: conditions — Recurrence

INTERVENTIONS:
Procedure: CO2 laser surgery
Procedure: ultrasonic surgical aspiration

SUMMARY:
1. To compare the recurrence rate between the use of laser vaporization and ultrasonic surgical aspiration in the treatment of vulvar and vaginal dysplasias
2. To compare healing related complications, post-operative pain, and scarring between the two procedures.

DETAILED DESCRIPTION:
First line of treatment for vulvar intraepithelial neoplasia (VIN) and vaginal intraepithelial neoplasia (VAIN) is not well defined. Laser vaporization and ultrasonic surgical aspiration are both accepted surgical modalities used in the treatment of vulvar and vaginal dysplasias, however no prospective study has been done to compare the two procedures. The specific aims of this research study include:

1. To compare the recurrence rate between the use of laser vaporization and ultrasonic surgical aspiration in the treatment of vulvar and vaginal dysplasias in a prospective, multi-institutional, randomized clinical trial.
2. To compare healing related complications, post-operative pain, and scarring between the two procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with vulvar or vaginal dysplasias or condylomas that require surgical intervention will be informed of the study by the treating physician
* Pre-operative biopsies to confirm presence of dysplasia / condyloma. Patients with dysplasias of grade 3 / CIS will be included at the discretion of the treating surgeon and will have had invasion confidently excluded by clinical exam and biopsy.

Exclusion Criteria:

* Patients under the age of eighteen or who are pregnant will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2005-12-31 (Actual); Study Completion 2005-12-31 (Actual)

PRIMARY OUTCOMES:
recurrence rate

SECONDARY OUTCOMES:
pain
side effects
complications

CONTACTS AND LOCATIONS:
Overall Officials: Vivian von Gruenigen, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Derived] von Gruenigen VE, Gibbons HE, Gibbins K, Jenison EL, Hopkins MP. Surgical treatments for vulvar and vaginal dysplasia: a randomized controlled trial. Obstet Gynecol. 2007 Apr;109(4):942-7. doi: 10.1097/01.AOG.0000258783.49564.5c. PMID 17400858